CLINICAL TRIAL: NCT06149429
Title: The Impact of a Novel Virtual Reality Protocol on Presence and Symptom Severity at the End-of-life.
Brief Title: Virtual Reality at End-of-life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: State University of New York - Upstate Medical University (Other)
Responsible Party: Principal Investigator, Catherine Mann, Clinical Professor, State University of New York at Buffalo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00007462
Record Dates: First submitted 2023-11-20; First posted 2023-11-29 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: End of Life; Pain; Nausea; Fatigue; Well-Being, Psychological; Depression; Dyspnea; Appetite Loss; Anxiety
Keywords: Hospice; Serious Illness; Virtual reality; End-of-life
MeSH Terms: conditions — Death; Pain; Nausea; Fatigue; Psychological Well-Being; Depression; Dyspnea; Anorexia; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Single group open pilot, pre- post-intervention study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single-Arm Open Pilot (Experimental): Pre- Post-intervention design. The intervention that participants will be experiencing is personalized virtual reality experiences. The content of this experience will be determined at the initial visit during which the participant will complete a preference questionnaire which identifies the location they want to "go" to. These experiences will be filmed on the insta360 One R camera by the research coordinator. Each experience will be approximately 20 minutes. To view the videos participants will wear the Oculus Quest 2 virtual reality headset.
  Interventions: Behavioral: Personalized virtual reality experience

INTERVENTIONS:
Behavioral: Personalized virtual reality experience — The intervention that participants will be experiencing is personalized virtual reality experiences. The content of this experience will be determined at the initial visit during which the participant will complete a preference questionnaire which identifies the location they want to "go" to. These experiences will be filmed on the insta360 One R camera by the research coordinator. Each experience will be approximately 20 minutes. To view the videos participants will wear the Oculus Quest 2 virtual reality headset.

SUMMARY:
The purpose of this research is to determine the effect that repeated, personalized virtual reality experiences have on symptom severity, comparing self-reported symptom severity both pre and post each session, and overtime across sessions. Researchers will also determine if this intervention results in a high rating of presence in VR, and if presence is related to the magnitude of the change in symptoms.

DETAILED DESCRIPTION:
The purpose of this research is to determine the effect that repeated, personalized virtual reality experiences have on symptom severity, comparing self-reported symptom severity both pre and post each session, and overtime across sessions. The researchers will also determine if this intervention results in a high rating of presence in VR, and if presence is related to the magnitude of the change in symptoms.

H1: Symptom severity will decrease from pre-intervention to post-intervention. H2: The change in symptom severity will be greater in session two than it was in session one.

H3: Presence score will be higher in session two than session one. To recruit 30-40 participants, the researchers will have the clinical team working to help the research team identify eligible participants from existing caseloads. Researchers will include all hospice eligible patients, this includes people who are enrolled in hospice care but also a subset of those who are enrolled in palliative care who qualify for hospice but have refused to or haven't yet transitioned to hospice care. The site serves about 670 (as of May 2023) patients a month. Therefore, it is the researcher's intent to recruit about 3 patents per month, or a total of 30-40 patients (about 5% of the monthly population) over the course of one year.

The intervention that participants will be experiencing is personalized virtual reality experiences. The content of this experience will be determined at the initial visit during which the participant will complete a preference questionnaire which identifies the location they want to "go" to. These experiences will be filmed on the insta360 One R camera by the research coordinator. Each experience will be approximately 20 minutes. To view the videos participants will wear the Oculus Quest 2 virtual reality headset.

ELIGIBILITY:
Healthy volunteers are not applicable to this study as they study focuses on pain and symptom management at end-of-life through the virtual reality experience.

Inclusion Criteria:

* Patients who are hospice care eligible as defined by the Medicare Hospice benefit and receive hospice or palliative care from Hospice and Palliative Care Buffalo.

Exclusion Criteria:

* Their Palliative Performance Score (PPS) is below 30.
* They are not cognitively intact (display symptoms of delirium or senility, or have a cognitive diagnosis such as Alzheimer's or Dementia) as measured by the Confusion Assessment Method (CAM) (Inouye et al., 1990)
* They have hearing, vision, or speech impairments that are uncorrected.
* They have current symptoms of or a history of dizziness, nausea, headaches, migraines, seizures, or motion sickness.
* They do not speak English.
* They are not 18 years old.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2023-10-23 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
Edmonton Symptom Assessment System - Revised (ESAS) | Two weeks
  End-of-life symptom assessment

SECONDARY OUTCOMES:
igroup presence questionnaire (IPQ) | Two weeks
  Presence during virtual reality experience

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Mann, EdD, Principal Investigator — SUNY Buffalo
Locations (1):
- Hospice and Palliative Care Buffalo, Cheektowaga, New York, United States

IPD SHARING:
Plan to Share IPD: No
Due to the sensitive nature of the study population at end-of-life and small sample size we feel that it poses undue risk for harm due to potential for anonymity being compromised.